CLINICAL TRIAL: NCT04459936
Title: A Multifactorial 'Urica Cor Intervention' to Prevent Cardiovascular Disease in People With Gout: Protocol for the Multicentre, Randomised Controlled, Blinded Endpoint URICORI Trial
Brief Title: Urica Cor Intervention (URICORI) Trial
Acronym: URICORI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been terminated due to inclusion difficulties during the worldwide Covid-19 pandemic.
Sponsor: Torkell Ellingsen (Other)
Collaborators: Odense University Hospital (Other); Frederiksberg University Hospital (Other); Oak Foundation (Other); The Danish Rheumatism Association (Other); Region of Southern Denmark (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Torkell Ellingsen, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OL10224607
Record Dates: First submitted 2020-05-17; First posted 2020-07-07 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Gout; Cardiovascular Diseases; Dyslipidemias; Hypertension; Diabetes; Behavior, Smoking
MeSH Terms: conditions — Gout; Cardiovascular Diseases; Dyslipidemias; Hypertension; Diabetes Mellitus; Smoking

STUDY DESIGN:
Intervention Model Description: The study is a randomised, open label, blinded endpoint trial, with balanced randomisation (1:1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Management by Rheumatologist (Experimental): Treatment of modifiable risk factors for cardiovascular disease managed by the Rheumatologist according to national guideline.
  Interventions: Other: URICORI
- Management by General Practitioner (Active Comparator): Treatment of modifiable risk factors for cardiovascular disease managed by the General Practitioner according to national guideline.
  Interventions: Other: CONTROL

INTERVENTIONS:
Other: URICORI — Treatment for cardiovascular risk factors according to national guideline administered at the department of Rheumatology
  Arms: Management by Rheumatologist
Other: CONTROL — Treatment for cardiovascular risk factors according to national guideline administered at the General Practitioner
  Arms: Management by General Practitioner

SUMMARY:
The objective of the Urica Cor Intervention (URICORI) trial is to evaluate the effectiveness of a one-year, intervention of modifiable risk factors for CVD administered in a rheumatology outpatient clinical setting, compared with conventional treatment for modifiable risk factors for CVD in people with gout.

DETAILED DESCRIPTION:
Introduction: Gout has been associated with a number of comorbidities including cardiovascular disease (CVD). Mounting evidence suggests that hyperuricaemia and gout are associated with a high risk for CVD. Gout is closely related to hypertension, dyslipidaemia, obesity and metabolic syndrome, all well-known factors contributing to the development of CVD. Gout management guidelines all agree that comorbidity screening is relevant and thus should be implemented in contemporary gout management. However, no specific strategy for management of CVD risk factors, in a gout population, exists.

Objective: The objective of the Urica Cor Intervention (URICORI) trial is to evaluate the effectiveness of a one-year, intervention of modifiable risk factors for CVD administered in a rheumatology outpatient clinical setting, compared with conventional treatment for modifiable risk factors for CVD in people with gout.

Design: The study is a randomised, open label, blinded endpoint trial, with balanced randomisation (1:1) conducted in four rheumatology outpatient clinics in Denmark. The investigators aim to recruit 266 people with gout, fulfilling the current EULAR ( European League against Rheumatism)/ ACR (American College of Rheumatology) gout classification criteria. Eligible patients will be randomised to receive either conventional (control group) treatment for CVD risk factors administered by their general practitioner according to national guidelines (NG) versus the URICORI programme, administered at the rheumatology department, targeting the same CVD risk factors according to NG. Both groups will be treated for gout at their local department of rheumatology.

End Points: primary end point is a composite endpoint. By inclusion in the URICORI programme all participants will be considered a member of one of four categories derived from the Systematic Coronary Risk Estimation (SCORE) screening programme designed to assess the 10 year risk of fatal cardiovascular disease in European low risk population. As a consequence, participants will be classified as responder after 12 months if all national treatment targets for LDL cholesterol, HbA1c, Blood pressure (systolic and diastolic), according to their SCORE risk profile, is met and no commencement of smoking. If not, participants will be classified as non-responders.

Key secondary end points: Change from baseline of LDL cholesterol, HbA1c, systolic blood pressure, diastolic blood pressure, smoking status and change from baseline in serum urate. Exploratory end points: Proportion of participants achieving treatment target for LDL cholesterol, HbA1c, systolic blood pressure, diastolic blood pressure, change in smoking status (commencement and cessation) and proportion of participants achieving serum urate < 36.0 mmol/l or serum urate < 0.30 mmol/l for tophaceous disease.

After year 1 and year 5, the first occurrence of any serious cardiovascular event (cardiovascular death, nonfatal myocardial infarction, nonfatal stroke or urgent revascularization due to unstable angina) during the URICORI trial will be registered. Death and hospitalisation during the URICORI trial will also be evaluated after year 5. Events will be determined by medical record review and evaluated by the endpoint adjudication committee. The Outcome Measures in Rheumatology (OMERACT) endorsed Core Domain Set for us in trials in gout will measured during and after the one-year URICORI intervention trial.

Ethics and dissemination: The local ethics committee in the region of southern Denmark and the Danish data agency in the region of southern Denmark will approve this protocol prior to commencement.

ELIGIBILITY:
Inclusion Criteria:

* Gout according to current EULAR/ACR (American College of Rheumatology) gout classification criteria
* Age >18 years
* Plasma LDL >3.0 mmol/L
* Agreeable to start treatment for CVD risk factors if indicated
* Ability to give informed consent
* Ability to communicate via telephone

Exclusion Criteria:

* Other inflammatory diseases requiring immunosuppressant therapy.
* Age >70 years.
* Active cancer (in active treatment).
* Chronic kidney disease (eGFR <30 ml/min/1.73m2).
* People whose behaviour or lifestyle would render them less likely to comply with the study protocol (i.e., abuse of alcohol, substance misuse or debilitating psychiatric conditions).
* Familial hypercholesterolemia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Responders (Dichotomised: responder/non-responder) | 1 year from inclusion
  Primary end point is a composite endpoint. By inclusion in the URICORI trial all participants will be considered a member of one of four categories derived from the Systematic Coronary Risk Estimation (SCORE - screening programme designed to assess the 10 year risk of fatal cardiovascular disease in European low risk population, range 0-24%). As a consequence, participants will be classified as responder after 12 months if all national treatment targets for LDL cholesterol, HbA1c, Blood pressure (systolic and diastolic), according to their SCORE risk profile, is met and no commencement of smoking. If not, participants will be classified as non-responders.

SECONDARY OUTCOMES:
LDL Cholesterol | 1 year from inclusion
  Change from baseline of LDL Cholesterol (mmol/L)
HbA1c | 1 year from inclusion
  Change from baseline of HbA1c (mmol/mol).
Systolic blood pressure | 1 year from inclusion
  Change from baseline Systolic blood pressure (mmHg).
Diastolic blood pressure Change from baseline Diastolic blood pressure (mmHg). | 1 year from inclusion
  Change from baseline Diastolic blood pressure (mmHg)
Smoking | 1 year from inclusion
  Change in smoking status (dichotomised yes/no)
Serum Urate | 1 year from inclusion
  Change from baseline in serum urate (mmol/L)

OTHER OUTCOMES:
LDL cholesterol | 1 and 5 years from inclusion
  Proportion of participants achieving treatment target for LDL cholesterol (mmol/L)
HbA1c | 1 and 5 years from inclusion
  Proportion of participants achieving HbA1c (mmol/mol) treatment target.
Systolic blood pressure | 1 and 5 years from inclusion
  Proportion of participants achieving treatment target for systolic blood pressure (mmHg)
Diastolic blood pressure | 1 and 5 years from inclusion
  Proportion of participants achieving treatment target for diastolic blood pressure (mmHg)
Smoking | 1 and 5 years from inclusion
  Proportion of participants with change in smoking status (commencement and cessation)
Serum urate | 1 and 5 years from inclusion
  Proportion of participants achieving serum urate < 36.0 mmol/l or if tophaceous disease serum urate < 0.30 mmol/l
Cardiovascular event | 1 year form inclusion
  Proportion of participants with any serious cardiovascular event during the first year of the URICORI trial.
Serious cardiovascular event | 5 years from inclusion
  Proportion of patients with any serious cardiovascular event during the 5-year URICORI trial. (serious cardiovascular event: cardiovascular death, non-fatal myocardial infarction, non-fatal stroke or urgent revascularization due to unstable angina)
Death | 5 years from inclusion
  Death from any cause (death will be classified as due to either cardiovascular or non-cardiovascular)
Hospitalisation | 5 years from inclusion
  Hospitalisation due to elective or acute cardiovascular reasons during the URICORI trial.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Morillon, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
If other research groups could benefit from the IPD (individual patient data ), the data will be shared after individual evaluation by the trial sponsor.

DOCUMENTS (1):
  • Study Protocol (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT04459936/Prot_000.pdf